CLINICAL TRIAL: NCT02258178
Title: Flucelvax Pregnancy Registry: an Observational Study on the Safety of Flucelvax Exposure in Pregnant Women and Their Offspring
Brief Title: Flucelvax Pregnancy Registry
Status: Withdrawn | Type: Observational
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Other Study IDs: V58_36OB
Record Dates: First submitted 2014-09-25; First posted 2014-10-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Pregnant Women, Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- 1, Flucelvax: Flucelvax exposure in pregnancy
  Interventions: Biological: Flucelvax (cTIV)

INTERVENTIONS:
Biological: Flucelvax (cTIV) — vaccine exposure in routine care (no vaccination per protocol)

SUMMARY:
The goal of the registry is to develop a better understanding of the safety of Flucelvax in women and their offspring who were exposed to the vaccine during pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy women pregnant women aged 18 years or older within the US who were immunized with the Flucelvax vaccine at any time during pregnancy.The registry will allow eligible pregnant women to selfenroll and also allow HCPs to report de-identified data on pregnancy exposures and outcomes.
* Sufficient evidence to confirm that Flucelvax exposure occurred during pregnancy
* Sufficient information to determine whether the pregnancy is prospectively or retrospectively registered (ie, whether the outcome of pregnancy was known at the time of first contact with the registry)
* Date the pregnancy exposure is registered
* Full reporter (ie, HCP) contact information to allow for follow-up (name, address,etc) The primary population for analysis will include prospectively enrolled pregnancies exposed to Flucelvax that are not lost to follow-up (ie, with outcome information that meet the minimum criteria for evaluation)

Exclusion Criteria:

* Invalid registry reports and pregnancies deemed lost to follow-up will be excluded from the primary analysis. Retrospective reports will not be included, although retrospective cases with MCMs will be reviewed and reported separately.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women aged 18 years or older within the US who were immunized with the Flucelvax vaccine at any time during pregnancy.The registry will allow eligible pregnant women to selfenroll and also allow HCPs to report de-identified data on pregnancy exposures and outcomes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
major congenital malformation | From time of enrollment during pregnancy to time of delivery or pregnancy termination
preterm birth | From time of enrollment during pregnancy to time of delivery or pregnancy termination
low birth weight | From time of enrollment during pregnancy to time of delivery or pregnancy termination

OTHER OUTCOMES:
Live birth | From time of enrollment during pregnancy to time of delivery or pregnancy termination
stillbirth | From time of enrollment during pregnancy to time of delivery or pregnancy termination
spontaneous abortion | From time of enrollment during pregnancy to time of delivery or pregnancy termination
ectopic pregnancy | From time of enrollment during pregnancy to time of delivery or pregnancy termination
molar pregnancy | From time of enrollment during pregnancy to time of delivery or pregnancy termination

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Wilmington, North Carolina, United States